CLINICAL TRIAL: NCT07055893
Title: Immunogenicity and Safety of a Rabies Vaccine (Serum-free Vero Cell), Freeze-dried in Comparison With Verorab®, in a Simulated Post-exposure Prophylaxis Regimen in Healthy Populations Aged ≥1 Years: A Randomized, Double-Blind, Active-controlled Phase Ⅲ Clinical Trial
Brief Title: Immunogenicity and Safety of Rabies Vaccine (Serum-free Vero Cell) in a Simulated Post-exposure Prophylaxis Regimen
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PVRV-sf-3002
Record Dates: First submitted 2025-05-27; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Rabies (Healthy Volunteers)
Keywords: rabies vaccine; Serum-free; post-exposure prophylaxis
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinovac rabies vaccine (Experimental): Participants will be randomly assigned to receive Sinovac rabies vaccine.
  Interventions: Biological: Rabies vaccine
- Sanofi Pasteur Verorab® (Active Comparator): Participants will be randomly assigned to receive the marketed rabies vaccine Verorab®
  Interventions: Biological: Verorab®

INTERVENTIONS:
Biological: Rabies vaccine — Receiving five doses of rabies vaccine manufactured by Sinovac using the "Essen" PEP schedule
  Arms: Sinovac rabies vaccine
Biological: Verorab® — Receiving five doses of marketed rabies vaccine manufactured by Sanofi using the "Essen" PEP schedule
  Arms: Sanofi Pasteur Verorab®

SUMMARY:
To demonstrate the immunogenicity of Sinovac rabies vaccine is non-inferior to the active-controlled rabies vaccine (Verorab®) after post-exposure prophylaxis (PEP) vaccination, and to confirm its satisfying safety profile in the pediatric and adult population in a PEP schedule

DETAILED DESCRIPTION:
This is a Phase Ⅲ, randomized, double-blind, active-controlled study. A total of 390 healthy participants aged ≥1 years old will be enrolled. All participants will be randomized at a 2:1 ratio to receive Sinovac rabies vaccine (Trial group) or Sanofi Pasteur Verorab® (Control group), in an Essen schedule of 5 doses at Day 0, Day 3, Day 7, Day 14, Day 28 through intramuscular route (IM) as a simulated rabies PEP.

Blood samples for immunogenicity assessment will be collected at Day 0, Day 14, Day 28, and Day 42. For safety assessment, the solicited local and systemic adverse events (AEs) within 7 days after each-dose vaccination (If the vaccination interval is less than 7 days, the actual interval shall prevail), as well as unsolicited AEs from the first-dose vaccination until 28 days after the last-dose vaccination will be actively monitored. Serious adverse events (SAEs) will also be collected during the whole study period.

ELIGIBILITY:
Inclusion Criteria:

1. Populations aged ≥1 years old;
2. Participants and/or participants' parents/legal guardians are able to understand and sign the informed consent form (ICF) voluntarily;
3. Participants are able to comply with the study procedures based on the investigator's assessment;
4. In a stable health status (defined as a stable preexisting disease status during the past 3 months, i.e., no change in treatment or hospitalization due to exacerbation of preexisting diseases);
5. Participants were tested negative for HIV, Syphilis, Hepatitis B, Hepatitis C infection at the screening of this study (the test result should be provided);
6. Female participants aged ≥15 years old with childbearing potential were tested negative for urine pregnancy test pre-vaccination, and also need to have effective contraceptive measures in the previous 2 weeks pre-vaccination.
7. Participants of childbearing potential and their partners are willing to take effective contraceptive measures and have no sperm or ovum donation plan from the time of signing ICF to 28 days after the last dose of vaccination;
8. Participants should provide verifiable identifications, and contact or be contacted with the investigators during the study period

Exclusion Criteria:

1. Fever on vaccination day, with axillary temperature >37.0°C (aged ≥5 years old) or >37.3°C (aged 1~4 years old) pre-vaccination;
2. Previous vaccination against rabies (in pre- or post-exposure regimen) with either trial vaccines or licensed vaccines;
3. Previous administration with rabies immunoglobulins or monoclonal antibodies;
4. Bite by, or exposure to a potentially rabid animal in the previous 12 months with category Ⅱ or Ⅲ exposures;
5. Female participants who are currently lactating or pregnant;
6. Known serious allergy to vaccines or vaccine ingredients, such as severe urticaria, anaphylactic shock, allergic laryngeal edema, allergic purpura, or known other serious adverse reactions to vaccine;
7. With severe congenital malformations or developmental disorders, genetic defects, severe malnutrition;
8. With autoimmune diseases, immunodeficiency diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid diseases, asplenia, functional asplenia, and HIV infection);
9. With poor controlled chronic illnesses or history of severe diseases, including but not limited to cardiovascular diseases, hematological disorders, liver and kidney diseases, digestive system disorders, respiratory diseases, malignancies, a history of major organ transplantation, drug-uncontrolled hypertension (only for participants aged ≥18 years old: with systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg), or any other disease or medical condition that the investigator believes could interfere with the trial results;
10. With current or past history of severe neurological diseases (epilepsy, convulsions or seizures [excluding history of febrile seizures]) or psychiatric disorders, or presence of a family history of psychiatric disorders;
11. With coagulation disorders (eg. factor deficiency, platelet disorders), or history of bleeding, hematoma, or bruising following intramuscular injections or venipuncture;
12. Receipt of ≥14 days of immunosuppressive or other immunomodulatory therapy (prednisone ≥2mg/kg/day, or its equivalent), cytotoxic therapy within 180 days prior to screening, or plans for such treatment in this study;
13. With long-term alcohol abuse [>14 drinks per week (1 drink =14 g 100% alcohol =360 mL beer, or 150 mL wine, or 45 mL distilled liquor/liquor)] or substance abuse (repeated and heavy use of narcotic drugs, psychotropic drugs, volatile organic solvents, etc.)
14. Receipt of blood products or immunoglobulins within 180 days prior to screening, or plans to receive these treatments in the study;
15. Receipt of other investigational drugs/vaccines within 30 days prior to screening, or plans to receive such drugs or vaccines during the study period;
16. Currently participating in other vaccine or drug clinical trials, or plan to participate in other clinical trials during the study;
17. Receipt of live-attenuated vaccines within 14 days prior to screening, or subunit or inactivated vaccines within 7 days prior to screening;
18. Presence of skin injuries, inflammation, ulcers, rashes, scars, or other conditions at the intended vaccination site that may interfere with drug administration or observation of local reactions;
19. Acute onset of various acute diseases or chronic diseases within the past 7 days, or known or suspected active infections;
20. Any other factors considered by the investigator to make the participant unsuitable for participation in the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving a rabies virus neutralizing antibody (RVNA) titer ≥0.5 IU/mL | Day 14 and Day 28 after the first dose vaccination

SECONDARY OUTCOMES:
Geometric mean concentrations (GMCs) of RVNA titers | Day 14, Day 28 and Day 42 after the first dose vaccination
Proportion of participants achieving a RVNA titer ≥0.5 IU/mL | Day 42 after the first dose vaccination
Incidence of adverse reactions | Up to 28 days after the last-dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ume Sughra, Dr., Principal Investigator — Director Research, Al-Shifa Research Centre; Professor of Public Health, Al-Shifa Trust Eye Hospital
Locations (1):
- Al-Shifa Trust Eye Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No